CLINICAL TRIAL: NCT01080001
Title: Impact of Fatigue in the Quality of Life of Patients With Multiple Sclerosis in Argentina
Brief Title: A Observational, Prospective Study to Assess the Impact of Fatigue in the Quality of Life of Patients With Multiple Sclerosis in Argentina
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200077-506
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Sclerosis, Relapsing-remitting
Keywords: Multiple sclerosis; Multiple sclerosis, Relapsing-remitting; Expanded Disability Status Scale; Fatigue; Hamilton Depression Inventory; Depression
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Fatigue; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an observational, non-controlled, multicentric, prospective study planned to be conducted in 66 subjects diagnosed with multiple sclerosis (MS) in 20 centres of Argentina. Fatigue is recognized as one of the most frequent symptoms of MS with a high incidence in MS subjects. The link between fatigue and the degree of disability and other manifestations of the disease, such as depression has not been yet clearly understood. Hence, this study aims to understand the way in which fatigue impairs the quality of life (QoL) of MS subjects. This epidemiologic study can contribute to a better understanding of the way in which fatigue correlates with depression and the intensity with which both situations impact on the QoL of MS subjects.

DETAILED DESCRIPTION:
Fatigue is recognized as one of the most frequent symptoms of MS and its impact on QoL of subjects is high. Fatigue in MS is sometimes considered as a prodromic symptom or as a peculiar symptom that must be differentiated from natural fatigue, pathological fatigue of other chronic diseases; as well as from fatigue caused by the excessive effort in case of gait disorder, spasticity or paresis. The origin of the fatigue symptom in MS is unknown and the cause is likely to be multifactorial. The evaluation of the fatigue is challenging, due to its variability and hence, scales such as Krupp's Fatigue Severity Scale (FSS) has been developed for measuring MS fatigue.

OBJECTIVES

Primary objective:

* To determine the impact of fatigue on QoL of MS subjects in Argentina

Secondary objective:

* To evaluate correlation between FSS and disability, depression, demographic variables; and between FSS and the use of disease modifying drugs
* To determine the impact of depression and neurological disability on QoL of MS subjects in Argentina

The subjects will be managed with the clinical and therapeutic elements that the treating doctor considers appropriate, without modifying their decisions due to the subject inclusion into the study. The epidemiologic data required by this study will be collected by the investigator from the documents in which each subject visit is registered, whether programmed or not. Once the recruiting period of 12 months is over, the collection of data will continue during the full 24 months period for each subject. The closure of the study will be marked by the follow-up of the last subject who entered the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with MS diagnosis (McDonald's criteria) in its relapsing remitting form
* Subjects between 21-60 years of age
* Subjects who did not have relapses during the 3 months before the inclusion
* Subjects with more than 1 year since the MS diagnosis or with a clinically defined MS

Exclusion Criteria:

* Subjects with life expectancy of less than 5 years at the moment of inclusion
* Subjects with other associated neurological disease
* Subjects with psychiatric diseases
* Subjects who have familiar antecedents (first grade) of severe depression
* Subjects with alcohol or drug abuse
* Subjects who are pregnant
* Subjects with FSS between 4 and 5
* Subjects who have used anxiolytics and anti depressants that could affect the fatigue symptoms during the 3 months before the inclusion

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects diagnosed with MS in Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis International Quality of Life (MusiQoL) in multiple sclerosis fatigue (MSF) [Fatigue Severity Scale (FSS) >5] versus multiple sclerosis nonfatigue (MSNF) (FSS <4) subjects | Each visit conducted from Day 0 (Initial visit) to the closure of the study (End visit at 24 month)

SECONDARY OUTCOMES:
Demographic characteristics | Initial visit (Day 0)
  Demographic and baseline variables include age, gender, race, baseline disease severity, sleep history, and baseline sleep assessments.
Duration of the disease | Initial visit (Day 0)
  Identifying the number of years since disease onset.
Treatment or treatment changes | Each visit conducted from Day 0 (Initial visit) to the closure of the study (End visit at 24 month)
  identifying the agents used for the treatment and the treatment duration.
Expanded Disability Status Scale (EDSS) | Each visit conducted from Day 0 (Initial visit) to the closure of the study (End visit at 24 month)
  EDSS >=3,5 disability and EDSS <=3,5 no disability
Hamilton Depression Inventory-17 (HDI-17) | Each visit conducted from Day 0 (Initial visit) to the closure of the study (End visit at 24 month)
Fatigue Severity Scale (FSS) | Each visit conducted from Day 0 (Initial visit) to the closure of the study (End visit at 24 month)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Norma Aydeé Deri, Principal Investigator — Hospital Fernandez, Buenos Aires, Argentina
Locations (1):
- Hospital Fernandez de Buenos Aires, Capital Federal, Buenos Aires, Argentina